CLINICAL TRIAL: NCT04084223
Title: Added Value of Early Collected Ultrasound As Compared to Clinical Evaluation to Predict Definite Clinical Outcome and Therapeutic Response in Rheumatoid Arthritis Patients Treated by JAK Inhibitors
Brief Title: JAKPOT (JAK Inhibitors and Predictors of Outcome in RheumaToid Arthritis)
Acronym: JAKPOT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slower pace of enrollments
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Centre Hospitalier Universitaire de Nīmes (Other); University Hospital, Clermont-Ferrand (Other); University Hospital, Bordeaux (Other); University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RECHMPL18_0241
Record Dates: First submitted 2019-07-18; First posted 2019-09-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Rheumatoid Arthritis
Keywords: JAK Inhibitors; Ultrasound; Patients Reported Outcomes (PROs); Disease activity; Predictors; Therapeutic response
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Active RA patients group (Experimental): 64 active RA patients (DAS28>3,2 AND presence of ≥2 US synovitis with Power-Doppler≥2) with an inadequate response to methotrexate (MTX) starting a treatment with JAKi (tofacitinib ou baricitinib) will be evaluated at baseline, 1, 3 and 6 months in 5 centres.
  A clinical joint assessment will be performed and CRP will be tested to calculate DAS28-CRP. Several PROs will be completed: RAPID3, HAQ, pain, and patient global assessment of disease activity on a VAS.
  An US exam on 40 joints and 12 tendons will be performed by an independent investigator, looking for synovitis and tenosynovitis with B-Mode and Power Doppler. A Global US score (GLOESS) will be collected at each visit.
  Interventions: Other: Ultrasound

INTERVENTIONS:
Other: Ultrasound — An Ultrasound exam (not performed in routine care) will be performed at Baseline, 1, 3 and 6 months for protocol.
  All patients will also have CRP dosage (for DAS28 assessment), RAPID-3 and PROs (performed in routine care but analyzed for the study).

SUMMARY:
Rheumatoid arthritis (RA) is a chronic, progressive autoimmune disease associated with inflammation and destruction of joints and systemic effects, which result in significant impact on patient's quality of life and function.

Sustained remission or low disease activity is the target to achieve in RA management. Ultrasound (US) is an imaging technique potentially helpful at several steps of the disease. A semi-quantitative (0-3) score of synovitis combining B-mode and Power Doppler abnormalities has been developed (GLOESS), and its responsiveness has been demonstrated. Patients Reported Outcomes (PROs) are important parameters in patient perceived health and are increasingly used in clinical practice. Prediction of therapeutic response to biological and targeted synthetic DMARDs remains a challenge for clinician, due to the potential adverse events and the cost of these drugs. To date, only few clinical and biological tools usable in clinical practice have a prognostic value. US or PRO could have added value for this purpose.

Objectives :

* To determine the predictive added value of the variation of an US score to the variation of the DAS28-CRP (C-Reactive Protein) at 1 month on clinical outcome (low disease activity i.e. DAS28-CRP≤3.2) at 6 months, or on therapeutic response at 3 months (EULAR good or moderate response (DAS)), in RA patients starting a treatment with JAK (Janus Kinase) inhibitors (JAKi).
* To determine the predictive added value of the variation several PROs to the variation of the DAS28-CRP at 1 month on clinical outcome (low disease activity i.e. DAS28-CRP≤3.2) at 6 months, or on therapeutic response at 3 months (EULAR good or moderate response (DAS)), in RA patients starting a treatment with JAKi.

DETAILED DESCRIPTION:
Ultrasound (US) is an imaging technique increasingly used in rheumatologic practice. US is a noninvasive, bedside, objective and sensitive tool for visualizing synovial inflammatory joint changes in RA that were not detected by conventional clinical examination. US has added value over clinical management of RA patients and is potentially helpful at several steps of the disease: early diagnosis of early arthritis, evaluation of disease activity, identification of poor prognostic RA, and possibly confirmation of remission status before tapering treatment. The potential role of this technique in the management of RA has been highlighted by the recent EULAR recommendations on how to use imaging in RA clinical practice. Nevertheless, only few studies have evaluated the value of US to predict clinical outcome and therapeutic response. In a Spanish longitudinal study including 42 early RA patients, the number and grade of Power-Doppler ultrasound (PDUS) synovitis were the best parameters correlated with disease activity at following visit. Since 2004, the OMERACT (Outcome Measures in Rheumatology) group has evaluated metric properties of US in RA. A semi-quantitative (0-3) score of synovitis combining B-mode and Power Doppler abnormalities was defined, the PDUS Global OMERACTEULAR Synovitis Score (GLOESS). This score recently demonstrated its responsiveness in a multicentre therapeutic trial of patients starting a treatment by abatacept, as soon as after one week of treatment. However, in this study, variation of this score until 4 months failed to demonstrate a correlation with clinical status or response as measured by DAS28-derived criteria at 6 months, suggesting that these tools evaluate different aspects of disease activity in RA and should be considered complementary in clinical practice, or maybe that DAS28 is not a sufficient stringent composite score. A similar semi-quantitative (0-3) score of tenosynovitis was developed and validated by the OMERACT. On the other hand, no study to date has demonstrated the responsiveness of this tenosynovitis score in RA. However, one study compared intra-muscular glucocorticoid or glucocorticoid administered in soft tissues and demonstrated that peri-tendinous infusions were more efficient at 3 months, both clinically and with US.

Patient-reported outcomes (PROs) are questionnaires used in clinical trials and daily care, with answers directly collected from patients. They allow the evaluation of domains that are often neglected (fatigue, quality of life, subjective disease activity, sleep disorders, etc). PROs are used as multifunctional criteria and therefore can be used as prognostic, therapeutic-evaluation or therapeutic-decision outcomes. Many studies have compared patient self-assessment and evaluation of disease activity by an experienced clinician to determine whether substituting patient assessment of disease activity is possible.

Clinical response during the first 3 months is associated with remission or low disease activity in the long term (6 to 12 months) in some studies. However, the real added value of US (or PRO) to predict medium or long term clinical outcome is not so well-known.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥18 years
* 2010 (American College of Rheumatology) ACR-EULAR classification criteria for RA for ≥3 months
* Inadequate response to MTX (or other csDMARD) for ≥3 months, at stable dosage for ≥1 month
* Active disease defined by DAS28>3,2 AND presence of ≥2 US synovitis with Power-Doppler≥2,
* Starting a treatment with JAKi (baricitinib or tofacitinib),
* Patients previously treated with biologic (stopped for inadequate response or safety) could be included. Biologics will be stopped before entering in the study: Abatacept and all TNF (tumor necrosis factor) inhibitors: no use within 4 weeks before baseline visit; Rituximab: no use within 6 months before baseline visit.
* Informed signed consent

Exclusion Criteria:

* Patient not treated before by MTX (or other csDMARD). Patients with a contraindication or in whom MTX was stopped due to safety issue could be included. Patients treated by MTX will have MTX during the follow-up, others will be treated by JAKi monotherapy,
* Patients with a contraindication to baricitinib or tofacitinib (current infection, recent attenuated vaccine injection, cancer <5 years…) or treated previously with baricitinib or tofacitinib,
* Patients treated by glucocorticoids ≥10 mg/day and unstable dosage for <1 month or with ≥1 glucocorticoids injection <1 month.
* RA with Steinbrocker class IV damage status
* General exclusion criteria (pregnancy, breast feeding…)
* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2024-09-24 (Actual); Study Completion 2024-09-24 (Actual)

PRIMARY OUTCOMES:
Disease activity | 6 months
  DAS28-CRP evaluated by an ultra-sound-blinded investigator (score calculated with number of painful articulations, synovitis, and C-Reactive Protein ; DAS28 result > 3,2 : moderately active rheumatoid arthritis)

SECONDARY OUTCOMES:
Disease activity | 1 month
  DAS28-CRP evaluated by a blinded investigator
Disease activity | 3 months
  DAS28-CRP evaluated by a blinded investigator
Ultra-sound activity | 1 month
  GLOESS-US evaluated by a blinded investigator
Ultra-sound activity | 3 months
  GLOESS-US evaluated by a blinded investigator
Ultra-sound activity | 6 months
  GLOESS-US evaluated by a blinded investigator
Patient Reported Outcomes: Health assessment (RAPID3) | up to 6 months
  Health assessment evaluated by RAPID3 questionnaire (Routine Assessment of Patient Index Data 3), a validated questionnaire assessing 3 domains : physical function, pain and disease activity. To calculate RAPID-3 scores, each of the 3 individual measures (Patient Global Activity on a visual analogic scale [VAS], pain [VAS] and function were scored from 0-10 for a total of 30. High scores represent the most altered health state. Cut-off value of disease activity were defined and validated: RAPID3 ≤3: Remission; RAPID3 between 3.1 and 6.0: Low disease activity; RAPID3 between 6,1 and 12: moderate disease activity; RAPID3 >12: high disease activity.
Patient Reported Outcomes: Health assessment (HAQ) | up to 6 months
  Health assessment evaluated by HAQ, a validated Health Assessment Questionnaire disability index for rhumatoid arthritis (score range from 0: no difficulties, to 3: patient disability)
Patient Reported Outcomes: pain | up to 6 months
  Pain evaluated by patient with VAS (visual analog scale) from 0 to 100
Patient Reported Outcomes: global health | up to 6 months
  Disease activity evaluated by patient with VAS (visual analog scale) from 0 to 100

CONTACTS AND LOCATIONS:
Overall Officials: Gaël MOUTERDE, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Rheumatology Department, Lapeyronie Hospital, Montpellier, France